CLINICAL TRIAL: NCT01058798
Title: The Role of Glycosyltransferases in the Oncogenesis of Neuroblastoma
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Wen-Ming Hsu, National Taiwan University Hospital
Other Study IDs: 200903079R
Record Dates: First submitted 2010-01-27; First posted 2010-01-29 (Estimated); Last update posted 2010-01-29 (Estimated); Status verified 2010-01

CONDITIONS: Neuroblastoma
Keywords: Neuroblastoma; B4GALNT3; Prognosis
MeSH Terms: conditions — Neuroblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Neuroblastoma (NB) is the most common malignant tumor of infancy. Approximately 60% of NB patients are clinically diagnosed as the stage IV disease and have a very poor prognosis with a 5-year survival rate of no more than 30%. The mechanism underlying the tumorigenesis of NB remains largely unclear. It has been suggested that the pathogenesis of NB is due to a failure of differentiation or apoptosis of the embryonic NB cells.

Well-regulated glycosylation is essential for the normal development of the nervous system. Altered expression of glycosyltransferases with resulting dysregulated glycosylation of neuroblastic cells might lead to the development of NB. The β1,4-N-acetylgalactosaminyltransferase III (B4GALNT3) exhibits GalNAc transferase activity to form the GalNAcβ1,4GlcNAc (LacdiNAc or LDN) structure. The Drosophila B4GALNTA, homolog of human B4GALNT3, has been suggested to regulate the neuronal development. By immunohistochemical studies, we demonstrated that the expression of B4GALNT3 correlated well with histological grade of differentiation in 87 NB tumor samples. In addition, positive B4GALNT3 expression predicted a favorable patient's outcome. These evidences suggest that the regulation of glycosyltransferases is critical for the development of NB.

To further explore the role of glycosyltransferases in the differentiation and development of NB, we propose a 3-year project with the following 3 major aims:

Aim Ⅰ: Clarifying the effects of B4GALNT3 on NB cell behavior in vitro and in vivo. For further understanding the effects of B4GALNT3 on NB cells, NB cells with stable overexpression of B4GALNT3 are to be selected. Then NB cell phenotype and behavior changes after overexpression of B4GALNT3 are evaluated by in vitro assays as well as by a nude mice xenograft model. In addition, the expression of B4GALNT3 will be suppressed by siRNA, then the response of NB cells to ATRA-induced differentiation is evaluated.

Aim Ⅱ: Clarifying the target proteins glycosylated by B4GALNT3 as well as their associated downstream pathways in vitro and in vivo. The possible proteins glycosylated by B4GALNT3 are evaluated by comparing differential protein expressions between B4GALNT3-transfected and mock-transfected NB cells using proteomics analysis. NB tumor samples with low and high B4GALNT3 expression levels are also subjected to proteomics analysis to explore the possible target proteins glycosylated by B4GALNT3 in vivo. After identifying the target proteins modified by B4GALNT3, the downstream pathways to affect NB cell differentiation will also be evaluated.

Aim Ⅲ: Clarifying whether B4GALNT4, a family member of B4GALNT, plays a similar role as B4GALNT3, as well as how the expression of these enzymes are controlled epigenetically in human NB cell lines and tumor samples. The expression levels of B4GALNT4 in human NB samples are evaluated by RT-PCR and immunohistochemistry. The methylation status of the promoter sites of both B4GALNT3 and B4GALNT4 are examined in various NB cell lines as well tumor samples. Furthermore, NB tumor samples exhibiting high and low B4GALNT levels are subjected to microRNA array.

Altogether, our studies will not only establish the functional role of the family of glycosyltransferases in the cell behavior of NB, but also illustrate how the expression of glycosyltransferases are regulated epigenetically and how the glycosyltransferases affect NB cell behavior. Therefore, our results might shed light to the oncogenesis of NB as well as target therapy of NB.

ELIGIBILITY:
Inclusion Criteria:

* Neuroblastoma patients with complete follow-up and sufficient samples for study

Exclusion Criteria:

* Neuroblastoma patients without complete follow-up or sufficient samples for study

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: From year 1990 to 2008, pediatric neuroblastoma patients treated at National University Hospital, Taiwan
Sampling Method: Non-Probability Sample
Dates: Start 2008-01; Primary Completion 2008-02 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Ming Hsu, M.D., Ph.D., Study Director — National Taiwan University Hospital